CLINICAL TRIAL: NCT00214604
Title: An 18-week, Randomized, Multicenter, Phase 3b, Double-blind, Crossover Study, Followed by an 18-week Open-Label Period to Evaluate the Efficacy & Safety of the Lipid-Regulating Agents, Rosuvastatin & Pravastatin in the Treatment of Subjects With Dysbetalipoproteinemia (Frederickson Type III Hyperlipoproteinemia)
Brief Title: Type III Dysbetalipoproteinemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: D3560C00071
Record Dates: First submitted 2005-09-21; First posted 2005-09-22 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Hyperlipoproteinemia Type III
MeSH Terms: conditions — Hyperlipoproteinemia Type III | interventions — Rosuvastatin Calcium; Pravastatin

INTERVENTIONS:
Drug: Rosuvastatin — 10mg
  Other Names: Crestor
Drug: rosuvastatin — 20mg
  Other Names: Crestor
Drug: pravastatin — 40mg
  Other Names: Pravachol

SUMMARY:
Evaluation of the efficacy of rosuvastatin 10mg, rosuvastatin 20mg and pravastatin 40mg in subjects with dysbetalipoproteinemia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of dysbetalipoproteinemia defined as VLDL-C/VLDL-TG mass ratio >0.35 at Visit 2 or the concurrence of mixed hyperlipidemia (fasting TC ≥ 200mg/dL, fasting TG ≥ 200mg/dL at Visits 2 and 3) and a genotype of ApoE published to be associated with dysbetalipoproteinemia

Exclusion Criteria:

* Use of cholesterol-lowering drugs, lipid lowering dietary supplements or food additives after Visit 1 except in accordance with the protocol as co-administered therapy (i.e., a fenofibrate) with rosuvastatin 40mg at Weeks 30 to 36; current active liver disease or hepatic dysfunction, serum CK ≥ 3 times ULN (unless explained by exercise) anytime during dietary period, serum creatinine > 2.0 mg/dL or a history of renal transplantation before the treatment phase, fasting triglyceride > 1000 mg/dL at any time during the dietary lead-in or a history of pancreatitis while on treatment for dysbetalipoproteinemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-02; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in non-HDL-C after 6 weeks of treatment at a given dose during the 18-week randomized crossover period.

SECONDARY OUTCOMES:
Efficacy of once daily treatment with rosuvastatin 10mg, rosuvastatin 20mg and provastatin 40mg in subjects with dysbetalipoproteinemia after 6 weeks of treatment at any given dose during the 18-week randomized crossover period.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Crestor Medical Sciences Director, MD, Study Director — AstraZeneca
Locations (2):
- Research Site, Oslo, Norway
- Research Site, Cape Town, South Africa